CLINICAL TRIAL: NCT03070379
Title: The Application of Topical Pharyngeal Anesthesia in the Esophagogastroduodenoscopy Under Sedation
Brief Title: Topical Pharyngeal Anesthesia in Sedated Esophagogastroduodenoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 307-TA
Record Dates: First submitted 2017-02-23; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Esophagogastroduodenoscopy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Topical lidocaine pharyngeal anesthesia was performed.
  Interventions: Procedure: Topical lidocaine pharyngeal anesthesia
- Control group (No Intervention): No topical lidocaine pharyngeal anesthesia was performed.

INTERVENTIONS:
Procedure: Topical lidocaine pharyngeal anesthesia — Topical pharyngeal anesthesia by lidocaine was administrated 4-5 min before propofol sedation in patients who underwent esophagogastroduodenoscopy.
  Arms: Experimental group

SUMMARY:
At recent, the number of patients who underwent sedated esophagogastroduodenoscopy has been on the increase. For such patients, whether topical pharyngeal anesthesia is needed remains to be controversial. European Society of Gastrointestinal Endoscopy, European Society of Gastroenterology and Endoscopy Nurses and Associates, and the European Society of Anaesthesiology Guideline for non-anesthesiologist administration of propofol for GI endoscopy have not made any recommendation, because the role of pharyngeal anesthesia during propofol sedation for upper digestive endoscopy has not been assessed. Our study aimed at investigating whether topical lidocaine pharyngeal anesthesia could benefit patients who underwent esophagogastroduodenoscopy under propofol sedation.

DETAILED DESCRIPTION:
Propofol sedation has been widely applied in endoscopic examinations. For such patients, whether lidocaine topical pharyngeal anesthesia should be administrated is still in doubt. Considering the fact that lidocaine anesthesia may cause airway narrowing and anaphylaxis, it is important to clarify the role of lidocaine topical pharyngeal anesthesia in esophagogastroduodenoscopy under propofol sedation. Our study could test whether lidocaine topical pharyngeal anesthesia should be performed in sedated esophagogastroduodenoscopy in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 Years
* Patients who have indications for esophagogastroduodenoscopy
* American Society of Anesthesiology risk class 1, 2 or 3

Exclusion Criteria:

* Patients <18 years
* Patients with thrombocytopenia (platelet count < 50,000/microL) or elevated International Normalized Ratio (INR > 1.5)
* Hemodynamic instability
* Pregnancy and lactation
* Patients who are unable or unwilling to give an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Immediate throat pain score | 1 day
  Immediate throat discomfort will be recorded, and pain score (0 no pain - 10 most painful) will be given by the patients.

SECONDARY OUTCOMES:
Throat discomfort 1 day after the procedure | 1 day
  All the patients will be followed up by telephone 1 day after the endoscopic examination. Throat Discomfort will be recorded.
Adverse events | 1 day
  All the adverse events during the sedated endoscopic examination will be recorded.
Satisfaction score | 1 day
  Patients will give a satisfaction score of 0 (unsatisfied) -10 (very satisfied) based on their own experience.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Liu, M.D., Ph.D., Principal Investigator — Department of gastroenterology,Affiliated Hospital to Academy of Military Medical Sciences
Locations (1):
- Affiliated Hospital to Academy of Military Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heuss LT, Hanhart A, Dell-Kuster S, Zdrnja K, Ortmann M, Beglinger C, Bucher HC, Degen L. Propofol sedation alone or in combination with pharyngeal lidocaine anesthesia for routine upper GI endoscopy: a randomized, double-blind, placebo-controlled, non-inferiority trial. Gastrointest Endosc. 2011 Dec;74(6):1207-14. doi: 10.1016/j.gie.2011.07.072. Epub 2011 Oct 13. PMID 22000794
- [Background] Dumonceau JM, Riphaus A, Aparicio JR, Beilenhoff U, Knape JT, Ortmann M, Paspatis G, Ponsioen CY, Racz I, Schreiber F, Vilmann P, Wehrmann T, Wientjes C, Walder B; NAAP Task Force Members. European Society of Gastrointestinal Endoscopy, European Society of Gastroenterology and Endoscopy Nurses and Associates, and the European Society of Anaesthesiology Guideline: Non-anesthesiologist administration of propofol for GI endoscopy. Endoscopy. 2010 Nov;42(11):960-74. doi: 10.1055/s-0030-1255728. Epub 2010 Nov 11. PMID 21072716
- [Derived] Sun X, Xu Y, Zhang X, Li A, Zhang H, Yang T, Liu Y. Topical pharyngeal anesthesia provides no additional benefit to propofol sedation for esophagogastroduodenoscopy: a randomized controlled double-blinded clinical trial. Sci Rep. 2018 Apr 27;8(1):6682. doi: 10.1038/s41598-018-25164-7. PMID 29703990